CLINICAL TRIAL: NCT04701346
Title: Dietary Sulfur Amino Acid Restriction, Energy Metabolism and Obesity
Brief Title: Sulfur Amino Acids, Energy Metabolism and Obesity
Acronym: STAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Charles University, Czech Republic (Other); Maastricht University (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Kathrine Vinknes, Researcher, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 310475
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Overweight and Obesity
Keywords: Methionine; Cysteine; Sulfur amino acids; Dietary intervention; Plant-based diet
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low SAA diet (Experimental): Dietary intervention
  Interventions: Other: Low SAA diet
- High SAA diet (Active Comparator): Dietary intervention
  Interventions: Other: High SAA diet

INTERVENTIONS:
Other: Low SAA diet — Diet with low content of methionine and cysteine
  Arms: Low SAA diet
Other: High SAA diet — Diet with high content of methionine and cysteine
  Arms: High SAA diet

SUMMARY:
The primary objective of the trial is to establish the effects of dietary sulfur amino acid (SAA) restriction on body weight, body composition and energy expenditure in humans.

DETAILED DESCRIPTION:
Dietary SAA restriction is an established model for increasing lifespan and improving metabolic health in animal studies. Data from human studies are limited.

In this study the investigators will perform an 8-week dietary intervention with SAA restriction to characterise the effects on several parameters related to metabolic health including body weight, body composition, energy expenditure, lipid profile and gene expression profiles in adipose tissue. The aim is to translate findings from previous animal experiments to humans

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with overweight and obesity (BMI 27-35 kg/m2)
* Waist circumference > 80 cm for women and > 94 cm for men

Exclusion Criteria:

* Smoking
* Presence of chronic disease
* Established co-morbidities
* Already on a vegan diet or have been the last month
* Pregnancy
* Breastfeeding the last 3 months
* Unstable body weight the last 3 months
* High intensity training > 3 times weekly

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | At baseline, 4 and 8 weeks
  Kilograms

SECONDARY OUTCOMES:
Changes in resting energy expenditure | At baseline, 4 and 8 weeks
  Kilocalories
Changes in substrate oxidation | At baseline, 4 and 8 weeks
  Respiratory quotient
Changes in body composition | At baseline, 4 and 8 weeks
  Fat mass (kilograms) and lean mass (kilograms)
Changes in plasma concentrations of SAA and related intermediates and compounds | At baseline, 4 and 8 weeks
  Sulfite, thiosulfate, rhodanide, sulfate, total aminothiols (homocysteine, cysteine, glutathione gamma-glutamylcysteine, cysteinylglycine, cysteamine), and fractions of total cysteine, total glutathione and total homocysteine, cystathionine, lanthionine, homolanthionine, taurine hypotaurine, sarcosine, hydrogen sulfide, S-adenosylmethionine and S-adenosylhomocysteine
Changes in urine concentrations of SAA and related intermediates and compounds | At baseline, 4 and 8 weeks
  Including sulfite, thiosulfate, rhodanide, sulfate, total aminothiols (homocysteine, cysteine, glutathione gamma-glutamylcysteine, cysteinylglycine, cysteamine)
Changes in concentrations of plasma lipid profile | At baseline, 4 and 8 weeks
  Fatty acids, total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, ApoA1, ApoB
Changes in plasma makers of insulin sensitivity | At baseline, 4 and 8 weeks
  Concentrations of glucose and insulin
Changes in plasma concentrations of adipokines and appetite hormones | At baseline, 4 and 8 weeks
  Leptin, adiponectin, gastrin, ghrelin, cholecystokinin (CCK), glucagon-like peptide (GLP-1), oxyntomodulin, gastric inhibitory peptide (GIP), peptide YY (PYY), and pancreatic peptide (PP).
Changes in gene expression | At baseline, 4 and 8 weeks
  mRNA of proteins involved in SAA metabolism, lipid and energy metabolism in leucocytes and subcutaneous white adipose tissue samples
Vitamin status | At baseline, 4 and 8 weeks
  Plasma concentrations of folate, B12 and methylmalonic acid (MMA)
Changes in biomarkers related to obesity and energy metabolism | At baseline, 4 and 8 weeks
  Untargeted analyses of plasma, serum and tissue concentrations
Changes in fibroblast growth factor 21 (FGF21) | At baseline, 4 and 8 weeks
  Serum concentrations
Nitrogen balance | At baseline, 4 and 8 weeks
  24 h-urine urea nitrogen
Changes in gut microbiota | At baseline, 4 and 8 weeks
  Sequencing of fecal samples
Changes in short chain fatty acids | At baseline, 4 and 8 weeks
  Fecal concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Dr Retterstøl, Prof. dr med, Study Director — University of Oslo
Locations (1):
- Centre for Clinical Nutrition, University of Oslo/Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
EU privacy regulations do not permit public sharing of IPD as long as the project is ongoing. Anonymized data can be shared after the project and biobank permissions end in 2030.
  The study protocol will be published.

REFERENCES:
- [Derived] Olsen T, Vinknes KJ, Barvikova K, Stolt E, Lee-Odegard S, Troensegaard H, Johannessen H, Elshorbagy A, Sokolova J, Krijt J, Krizkova M, Ditroi T, Nagy P, Ovrebo B, Refsum H, Thoresen M, Retterstol K, Kozich V. Dietary sulfur amino acid restriction in humans with overweight and obesity: Evidence of an altered plasma and urine sulfurome, and a novel metabolic signature that correlates with loss of fat mass and adipose tissue gene expression. Redox Biol. 2024 Jul;73:103192. doi: 10.1016/j.redox.2024.103192. Epub 2024 May 17. PMID 38776754
- [Derived] Olsen T, Stolt E, Ovrebo B, Elshorbagy A, Tore EC, Lee-Odegard S, Troensegaard H, Johannessen H, Doeland B, Vo AAD, Dahl AF, Svendsen K, Thoresen M, Refsum H, Rising R, Barvikova K, van Greevenbroek M, Kozich V, Retterstol K, Vinknes KJ. Dietary sulfur amino acid restriction in humans with overweight and obesity: a translational randomized controlled trial. J Transl Med. 2024 Jan 9;22(1):40. doi: 10.1186/s12967-023-04833-w. PMID 38195568
- [Derived] Stolt E, Olsen T, Elshorbagy A, Kozich V, van Greevenbroek M, Ovrebo B, Thoresen M, Refsum H, Retterstol K, Vinknes KJ. Sulfur amino acid restriction, energy metabolism and obesity: a study protocol of an 8-week randomized controlled dietary intervention with whole foods and amino acid supplements. J Transl Med. 2021 Apr 15;19(1):153. doi: 10.1186/s12967-021-02824-3. PMID 33858441